CLINICAL TRIAL: NCT06581887
Title: Defining Outcome Measures for Behavioural and Emotional Problems in Dystrophinopathies
Acronym: D-BRAIN
Status: Recruiting | Type: Observational
Sponsor: University College, London (Other)
Collaborators: Sarepta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 21/WM/0267; 302390 (Other: IRAS)
Record Dates: First submitted 2024-08-08; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: DMD; BMD
Keywords: Antisense oligonucleotide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cohort: * Social Responsiveness Scale (SRS - II)
  * ADHD Rating scale (5th edition) (ADHD - RS V)
  * Child Behaviour Checklist (CBCL)
  * Revised Children's Anxiety and Depression Scale (RCADS-P)
  * Behaviour Rating Inventory of Executive Function (BRIEF - P)
  * Wechsler Intelligence test for children version V (WISC-V)
  * Autism Diagnostic Observation Schedule (ADOS)
  * Behavioural Assessment of the Dysexecutive Syndrome for Children (BADS-C)
  * Psychophysiological task: A task previously used to measure the emotional response of patients through the usage of visual and auditory aversive stimuli. The emotional response will be measured through skin conductance, heartrate, pupil responses.
  * Purdue Pegboard
  * A subset of patients will be also asked to undergo an MRI brain scan
  Interventions: Behavioral: Classical conditioning task

INTERVENTIONS:
Behavioral: Classical conditioning task — To evaluate the neurophysiological and physiological response to a classical conditioning task, which is comparable to findings that have been made in the mdx dystrophic mouse (deficient in Dp427). The investigators will assess correlations between the specific DMD/BMD genotype and susceptibility to conditioning, as well as the relationship between conditioning and behavioural/emotional characteristics of the syndrome.

SUMMARY:
Study aims to develop and to evaluate the neurophysiological and physiological response to a classical conditioning task.To better understand how Duchenne Muscular Dystrophy (DMD) and Becker Muscular Dystrophy (BMD) impacts mental health and how to assess it. Participants invited to complete questionnaires about behaviour, cognitive function and social interactions, complete computer tasks and have an optional MRI brain scan,

DETAILED DESCRIPTION:
The investigation aims to develop and to evaluate the neurophysiological and physiological response to a classical conditioning task, which is comparable to findings that have been made in the mdx dystrophic mouse (deficient in Dp427). The investigators will assess correlations between the specific DMD/BMD genotype and susceptibility to conditioning, as well as the relationship between conditioning and behavioural/emotional characteristics of the syndrome. At the end of the study, the objective is to deliver a comprehensive test battery that is suitable for use in a trial of AON delivery to improve brain function.

ELIGIBILITY:
Inclusion Criteria:

* DMD patients:

  1. Male
  2. Age range 7-17 years
  3. A genetically proven diagnosis of DMD.
  4. A genetic mutation that abrogates expression of Dp427 alone (assigned in DMD Group 1: Dp427-/Dp140+) or both Dp427 and Dp140 (assigned to DMD Group 2: Dp427-/Dp140-).
  5. Ability to consent/assent

BMD patients:

1. Male
2. Age range 7-17 years
3. A genetically proven diagnosis of BMD.
4. A genetic mutation that decreases expression of Dp427 alone (assigned to BMD Group 1), of both Dp427 and Dp140 (assigned to BMD Group 2).
5. Ability to consent/assent

Control participants:

1. Male
2. Age range 7-17 years.
3. Ability to consent/assent

Exclusion Criteria:

* DMD & BMD patients:

  1. Significant visual or hearing impairment
  2. Specific phobias or sensory sensitivities to stimuli similar to the ones used in this study
  3. Current participation in a clinical trial investigating a new drug involved in dystrophin modulation.
  4. Inability to consent (for parents/guardians or self-reporting participants aged 16 and 17) or assent. This will exclude the rare individuals with extremely severe learning disability, as the assent in these patients is impossible (or the consent in self-reporting participants aged 16 and 17).

Control participants:

1. Significant visual or hearing impairment
2. Specific phobias or sensory sensitivities to stimuli similar to the ones used in this study
3. Any diagnosis of neurological or psychiatric condition

General exclusion criteria for MRI:

1. Claustrophobia
2. Pacemakers and defibrillators
3. Nerve stimulators
4. Intracranial clips
5. Intraorbital or intraocular metallic fragments
6. Cochlear implants
7. Ferromagnetic implants (e.g. thoracic implant for scoliosis)
8. Inability to lie supine during less than 45 minutes
9. Not having a general practitioner
10. Severe learning disability which will require a general anaesthetic

Ages: 7 Years to 17 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Male
Study Population: 40 DMD, 30 BMD patients and 30 age-matched controls.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-09-13 (Actual); Primary Completion 2024-11-19 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Group differences between DMD, BMD and controls in the initial aversive unconditioned stimulus. | through study completion, an average of 2 years
  Following an emotional response task, an interim analysis will be done after the first 30 patients have been tested (10 DMD, 10 BMD, 10 controls). A favourable outcome will demonstrate a difference in the emotional response of these groups. Groups will complete questionnaires, an emotional response task, and a fine motor assessment.

SECONDARY OUTCOMES:
To observe any difference between and within BMD, DMD and control groups in regard to learning, habituation and extinction | through study completion, an average of 2 years
  This will be measured by analysis measuring any difference between and within groups (10 BMD, 10 DMD and 10 control). Physiological responses generated by the task will be measured, along with neural imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Muntoni, Professor, Principal Investigator — University College, London
Locations (1):
- UCL GOS Institute of Child Health, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The results of the study will be published in peer-reviewed scientific journal(s), presented at relevant national and international meetings, and reported as part of submissions to regulatory and funding bodies (Joint Research & Development Office, GOSH & ICH; NHS Research Ethics Committee; GOSH Charity). Participants will be asked if they wish to be contacted when the results are published, and if in agreement they will be informed by letter/email of any resulting publications.

REFERENCES:
- See also: Duchenne clinical trial listing — https://dmdhub.org/trials/d-brain/
- See also: Health Research Authority research summary — https://www.hra.nhs.uk/planning-and-improving-research/application-summaries/research-summaries/d-brain/